CLINICAL TRIAL: NCT06380582
Title: Indoor Air Quality, Temperature and Cognitive Performance
Acronym: AEOLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL85595.068.23
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-06

CONDITIONS: Indoor Air Quality; Temperature; Cognitive Performance
Keywords: Indoor air quality; Temperature; Cognition; Metabolism
MeSH Terms: interventions — Temperature

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Air flow (Experimental): low airflow and high airflow
  Interventions: Other: Temperature and Airflow combination
- Temperature (Experimental): 23C 40%RH or 35C 40%RH
  Interventions: Other: Temperature and Airflow combination

INTERVENTIONS:
Other: Temperature and Airflow combination — 23C 40%Relative Humidity (RH) low airflow, 23C 40%RH high airflow, 35C 40%RH low airflow, 35C 40% high airflow

SUMMARY:
Study design: A cross-over single-blinded treatment design will be used. Participants will undergo 4 different conditions: (1) low air flow and 23°C, (2) low air flow and 35°C, (3) high air flow and 23°C, and (4) high air flow and 35°C. Participants will be blinded to the air quality level; however, it is not possible to blind them to the temperature condition, as they will be able to perceive it as different.

Study population: The population consists of healthy young and middle-aged adults of both sexes between 18 and 40 years.

Intervention (if applicable): Each participant undergoes 4 conditions in randomized order. Two conditions consist of poor air quality defined as 3,000 ppm carbon dioxide and 23°C or 35°C temperature, respectively.

DETAILED DESCRIPTION:
Objective: This study aims to examine the effect of indoor air quality and temperature on human cognitive performance. The main research objective of this study is to examine how indoor air quality and temperature affects cognitive performance, respectively. As a secondary objective, it will be examined if a higher temperature of 35°C compared to 23°C amplifies the negative effect of low air flow vs. high air flow on cognitive performance. It will also be examined if human perceive the air quality as less pleasant under the higher temperature, even if the air quality itself does not change in terms of carbon dioxide concentration. Also, the physiological reaction towards poor air quality and elevated temperature will be examined in isolation and interaction.

Main study parameters/endpoints: The main study parameters are the achieved scores of the cognition test, mainly derived from the Cambridge Neuropsychological Test Automated Battery (CANTAB) and the Cognitive Ability Task. As secondary outcome, the physiological response will be examined. Specifically, it will be investigated how the air quality and temperature affect the following physiological parameters: Capillary blood CO2 and pH level, salivary cortisol and a-amylase and serum cytokine response, lung function, heart rate, respiration rate, skin temperature, core temperature, blood pressure, physical activity, and metabolic rate.

Primary Objective: The main research objective of this study is to examine how poor indoor air quality in terms of low air flow compared to high air flow and elevated temperature of 35°C compared to 23°C affect cognitive performance, respectively.

Secondary Objective(s): The following secondary objectives will be investigated in this study:

1. It will be examined whether the decline in cognitive performance is greater when low air quality to high air quality compared to when temperature levels are increasing from 23°C to 35°C.
2. It will be examined whether a higher temperature of 35°C compared to 23°C amplifies the negative effect of poor air quality.
3. It will be examined whether participants perceive the air quality as less satisfactory if temperature levels are higher indoors, even when the air quality is unchanged. It will be also examined to which physiological reactions poor air quality and elevated temperature lead. Specifically, the following objectives will be investigated:
4. It will be examined whether metabolic rate is affected under poor air quality conditions or higher temperature indicated by a change in CO2 production and oxygen consumption.
5. It will be examined whether poor air quality or higher temperature levels are associated with a stress response defined by a higher heart rate, higher respiration rate, higher blood pressure, higher alpha-amylase and cortisol levels, and a higher rate of non-exercise activity thermogenesis through increased physical activity.
6. It will be examined whether lung function in terms of forced expiratory volume and forced vital capacity are reduced when participants are exposed to poor air quality in combination with a higher temperature of 35°C.
7. It will be examined whether blood capillary carbon dioxide concentration and blood pH level are elevated under worse air quality in combination with a higher temperature of 35°C.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 to 40 years old
* Western-European background
* Generally healthy
* No medication which may influence the outcome parameters. This will be determined on a case-by-case basis. Contraceptive uses for women are allowed and will be verified through a questionnaire.
* Non-smokers or persons who quit smoking more than five years ago

Exclusion Criteria:

Participants, who do not want to be informed about unexpected medical findings, or do not wish that their treating physician will be informed, cannot participate in this study

* Individuals with a diagnosed physical or mental disability or attention deficit hyperactivity disorder (ADHD) or depression
* Any medication or medical condition that might interfere with the physiological outcome parameters or in some regards impair cognition
* Unstable body weight (weight gain or loss >3kg in the past three months)
* Participation in another biomedical study within 1 month prior to screening visit
* Shift workers
* Colour blindness
* Pregnancy
* People with a low haemoglobin or haematocrit concentration
* Not having visited or resided in a warm country in the last 3 months
* Participants with asthma or restricted lung function due to allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Cognition Morning | 1 month
  Cambridge Neuropsychological Test Automated Battery (CANTAB) once at 11am and once at 230pm
Cognition Afternoon | 1 month
  Cognitive Ability Task - once at 4pm

SECONDARY OUTCOMES:
Heart Rate (bpm) | 1 month
  Using a wearable heart rate belt for beat by beat
Metabolic Rate (ml/kg/min) | 1 month
  Omnical system with a minute frequency
Blood Pressure (mmHg) | 1 month
  Using an automate blood pressure cuff every hour
Blood samples | 1 month
  Blood drawn for future analysis 4 times every 2 hours
Saliva samples | 1 month
  Saliva collected for future analysis 4 times every 2 hours
Breathing rate | 1 month
  Spirometer used 4 times every 2 hours

OTHER OUTCOMES:
Temperature (C) | 1 month
  Room temperature using an environmental sensor
Humidity % | 1 month
  Relative Humidity using an environmental sensor
Carbon dioxide (CO2) concentration (ppm) | 1 month
  Carbon dioxide using an environmental sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Open Access upon request of fully anonymized data after initial analysis
Supporting Information: Study Protocol, SAP
Time Frame: Open Access upon request of fully anonymized data after initial analysis